CLINICAL TRIAL: NCT06028100
Title: The Effect of an Ultrasound-guided Sacral Erector Spinae Plane Block on the Post-operative Pain of Lumbar Discectomy Surgery
Brief Title: Sacral Erector Spinae Plane Block(ESPB) in Lumbar Discectomy
Acronym: ESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilge Olgun Keles (Other)
Responsible Party: Sponsor-Investigator, Bilge Olgun Keles, Assistant professor, Giresun University
Organization: Giresun University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/06
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Pain Management
Keywords: regional block; erector spinae plane block; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: 54 patients were included in the study, divided into two groups of 27 patients as esp block (group 1) and control group (group 2), both groups underwent standard general anaesthesia. The blocks were performed in the operating theatre at the end of the operation, before the patient woke up.A patient-controlled analgesia (PCA) device was given to both groups by another doctor blinded to the group, and Visual Analogue Scale (VAS) scores assessed for 24 hours.And total consumption of analgesic and rescue analgesics were recorded.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient did not know what was done to him/her because the block was performed before the patient woke up.
  The investigator who questioned postoperative pain and opioid consumption did not know to whom the block was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- espb group (Active Comparator): The first group underwent sacral espb at the end of surgery. The lumbosacral region was sterilised with povidine iodine and then draped with the patient in prone position. The linear ultrasound probe was placed in the midline on the spinous process of the 5th lumbar vertebra after the sterile covering had been applied. After observation of the sacrum, the level of the 2nd median crest was determined and the ultrasound probe was moved 1.5-2 cm laterally and the 2nd intermediate crest and the erector spinae muscle between the two were observed. 22 G 50 mm needle was advanced from caudal to cranial direction to the sacral crest using in-plane technique, after confirming the needle position with 1-2 ml saline, 0.25% bupivacaine 20 ml was administered, local anaesthesia was observed to spread cauda-cranially separating the erector spinae muscle from the sacral crest, the same procedure was performed on the opposite side
  Interventions: Procedure: sacral erector spinae plane block
- control group (No Intervention): The second group had no any block

INTERVENTIONS:
Procedure: sacral erector spinae plane block — espb from bilateral sacral level 2 with 20 ml %0,25 bupivacaine
  Arms: espb group

SUMMARY:
Several studies have shown that sacral espb blocks the dorsal ramus of spinal nerves. In lumbar discectomy operations, innervation of all tissues where pain occurs is provided by the dorsal ramus of the nerves. Based on this information, it was thought that sacral espb would be effective in lumbar discectomies. The investigators wanted to look at the effects of sacral erector spinae plane block on postoperative pain and opioid consumption in lumbar discectomy operations. There is no randomised controlled study on sacral espb in the literature. The researchers think that the results of the study are promising. Sacral espb is an easy-to-administer block with a low risk of complications and can be used effectively in lumbar discectomy analgesia.

DETAILED DESCRIPTION:
This prospective, randomised, controlled, double-blind, single-centre study was approved by our Ethics Committee (KAEK2023/06). The investigators followed the Consolidated Reporting Trials Standards (CONSORT). It was conducted in patients undergoing elective lumbar discectomy, and informed consent was obtained from the patients. They were randomised using a closed envelope technique, opened by the physician performing the block. 54 patients were included in the study, divided into two groups of 27 patients as esp block (group 1) and control group (group 2), both groups underwent standard general anaesthesia. The blocks were performed in the operating theatre at the end of the operation, before the patient woke up. The patients were unaware that the block was being performed on them. A patient-controlled analgesia (PCA) device was given to both groups by another doctor blinded to the group, and Visual Analogue Scale (VAS) scores assessed for 24 hours.

Standard monitoring (peripheral oxygen saturation, electrocardiogram, non-invasive arterial blood pressure monitoring) was performed. Anaesthesia induction was achieved with 1 mcg/kg fentanyl, 2 mg/kg propofol, 0.6 mg/kg rocuronium, and anaesthesia maintenance with 2% sevoflurane, 4 lt/min 50%/50% oxygen/nitrogen mixture. Both groups received 1 g IV paracetamol towards the end of surgery. The patients were extubated after 2 mg/kg of sugammadex and were transferred to the recovery room.

The first group underwent sacral espb at the end of surgery. The lumbosacral region was sterilised with povidine iodine and then draped with the patient in prone position. The linear ultrasound probe was placed in the midline on the spinous process of the 5th lumbar vertebra after the sterile covering had been applied. After observation of the sacrum, the level of the 2nd median crest was determined and the ultrasound probe was moved 1.5-2 cm laterally and the 2nd intermediate crest and the erector spinae muscle between the two were observed. 22 G 50 mm needle was advanced from caudal to cranial direction to the sacral crest using in-plane technique, after confirming the needle position with 1-2 ml saline, 0.25% bupivacaine 20 ml was administered, local anaesthesia was observed to spread cauda-cranially separating the erector spinae muscle from the sacral crest, the same procedure was performed on the opposite side.

All patient demographics, age, weight, and duration of surgery, post-operative VAS scores, blood pressure, heart rate and oxygen saturation values at 30 min, 1, 6, 12 and 24 hours, total tramadol consumption, rescue analgesic use, time of first rescue analgesic requirement, patient satisfaction and side effects were recorded.

The Shapiro-Wilk test was used to examine the normality of quantitative data. Comparison of normally distributed data was performed by independent samples t-test, and comparison of non-normally distributed data was performed by Mann-Whitney U test. Comparison of qualitative data was performed using the Pearson chi-squared test. Data were presented as mean ± standard deviation, median (minimum - maximum) and n (%). Statistical significance was accepted as p<0.05. In a previous study (9), the power analysis performed to detect a difference of 15.4 mg between the 48-hour opioid consumption values of the two groups (p<0.05) was calculated with 90% power and an effect size of 0.96, and the required sample size was determined to be 24 for each group. If 10-15% of patients were excluded from the study, 27 patients were included for each group and 54 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age,
* American Society of Anesthesiology(ASA) status 1-3 group

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients with known neuromuscular and haematological diseases
* Allergy to local anaesthetics
* Contraindications to regional anaesthesia
* Anatomical changes in the lumbo-sacral region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Patient pain scores | 24 hours
  Visual Analog Scala (0:No pain 10: Worst pain possible)
Patient total opioid consumption | 24 hours
  The number of patient controlled analgesia device boluses doses

SECONDARY OUTCOMES:
Nausea-vomiting | 24 hours
  The incidence of side effects described yes or no
Patient satisfaction | 24. hours
  Patient satisfaction (0:Not satisfied 10:Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Olgun Keleş, M.D., Study Director — Giresun University
Locations (1):
- Giresun Research and Training Hospital, Merkez, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since it is the first study on this subject in the literature

REFERENCES:
- [Result] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Result] Bajwa SJ, Haldar R. Pain management following spinal surgeries: An appraisal of the available options. J Craniovertebr Junction Spine. 2015 Jul-Sep;6(3):105-10. doi: 10.4103/0974-8237.161589. PMID 26288544
- [Result] Kilicaslan A, Aydin A, Kekec AF, Ahiskalioglu A. Sacral erector spinae plane block provides effective postoperative analgesia for pelvic and sacral fracture surgery. J Clin Anesth. 2020 May;61:109674. doi: 10.1016/j.jclinane.2019.109674. Epub 2019 Dec 4. No abstract available. PMID 31812367
- [Result] Chakraborty A, Chakraborty S, Sen S, Bhatacharya T, Khemka R. Modification of the sacral erector spinae plane block using an ultrasound-guided sacral foramen injection: dermatomal distribution and radiocontrast study. Anaesthesia. 2021 Nov;76(11):1538-1539. doi: 10.1111/anae.15549. Epub 2021 Jul 26. No abstract available. PMID 34309009
- [Result] Mistry T, Sonawane K, Balasubramanian S, Balavenkatasubramanian J, Goel VK. Ultrasound-guided sacral multifidus plane block for sacral spine surgery: A case report. Saudi J Anaesth. 2022 Apr-Jun;16(2):236-239. doi: 10.4103/sja.sja_723_21. Epub 2022 Mar 17. PMID 35431750